CLINICAL TRIAL: NCT04094805
Title: A Multicenter Randomized Open-label Clinical Trial of Vitamin D Combined With HD-DXM Versus HD-DXM for the Treatment of ITP
Brief Title: A Multicenter Randomized Study of Vitamin D Combined With HD-DXM Versus HD-DXM for the Treatment of ITP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITP-Vitamin D+HD-DXM
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Calcitriol; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rocaltrol Combining HD-DXM (Active Comparator): Rocaltrol 0.25 μg once per day, 1 month; HD-DXM (orally at 40 mg daily for 4d )
  Interventions: Drug: Rocaltrol; Drug: Dexamethasone
- HD-DXM (Active Comparator): HD-DXM (orally at 40 mg daily for 4d )
  Interventions: Drug: Rocaltrol

INTERVENTIONS:
Drug: Rocaltrol — Rocaltrol 0.25 μg daily for 1 month; HD-DXM (orally at 40 mg daily for 4d )
  Other Names: Calcitriol Soft Capsules
Drug: Dexamethasone — HD-DXM (orally at 40 mg daily for 4d )
  Arms: Rocaltrol Combining HD-DXM

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University in China. In order to report the efficacy and safety of vitamin D combining with high-dose dexamethasone for the treatment of adults with newly-diagnosed primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators anticipate to undertaking a prospective, multicenter, randomised controlled trial of 60 ITP adult patients. One part of the participants are randomly selected to receive vitamin D (given Rocaltrol orally at a dose of 0.25 μg per day for 1 month), combining with dexamethasone (given orally at a dose of 40 mg per day for 4 days, two-cycles with an interval of 10 days); the others are selected to receive high-dose of dexamethasone treatment plus placebo. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Serum calcium and creatinine are monitored. Adverse events are also recorded throughout the study. In order to report the efficacy and safety of vitamin D combining with high-dose dexamethasone therapy for the treatment of adults with ITP.

ELIGIBILITY:
Inclusion Criteria:

1. Corresponding to the diagnostic criteria for immune thrombocytopenia
2. Newly diagnosed ITP patients
3. To show a platelet count <30 * 10^9/L, and with bleeding manifestations
4. Willing and able to sign written informed consent

Exclusion Criteria:

1. Suffered from diseases associated with hypercalcemia.
2. Vitamin D intoxication
3. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit;
4. Received second-line ITP-specific treatments (eg, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) within 3 months before the screening visit; 3.Received high-dose steroids or IVIG in the 3 weeks prior to the start of the study;
5. Current HIV infection;
6. Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
7. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period;
8. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test;
9. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Sustained response to ITP treatments | 3 months after treatment started
  Percentage of patients maintaining PLT count over 30*10^9 without bleeding

SECONDARY OUTCOMES:
Evaluation of platelet response | 3 months after treatment started
  Complete response (CR)： A platelet count ≥ 100 * 10^9/L measured on two occasions > 7 days apart and the absence of bleeding.
  Response (R)： A platelet count ≥ 30 * 10^9/L and a greater than two fold increase in platelet count from baseline measured on two occasions > 7 days apart and the absence of bleeding.
  No response (NR)： A platelet count < 30 * 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No